CLINICAL TRIAL: NCT05548387
Title: A Randomized, Open Label, Single Dose, 4-period Replicate Crossover Clinical Trial to Evaluate the Pharmacokinetic Characteristics and Safety After Administration of a Fixed-dose Combination Drug of HCP2202 or Co-administration of RLD2202 and RLD2203 in Healthy Volunteers Under Fasting Conditions
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between HCP2202 and Co-administration of Each Component in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-SARA-102
Record Dates: First submitted 2022-09-06; First posted 2022-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: RLD2202 +RLD2203 Period 2: HCP2202 Period 3: RLD2202 +RLD2203 Period 4: HCP2202
  Interventions: Drug: HCP2202; Drug: RLD2202; Drug: RLD2203
- Sequence 2 (Experimental): Period 1: HCP2202 Period 2: RLD2202 +RLD2203 Period 3: HCP2202 Period 4: RLD2202 +RLD2203
  Interventions: Drug: HCP2202; Drug: RLD2202; Drug: RLD2203

INTERVENTIONS:
Drug: HCP2202 — Take it once per period.
Drug: RLD2202 — Take it once per period.
Drug: RLD2203 — Take it once per period.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety between HCP2202 and co-administration of each component in fasting condition in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~54 years in healthy volunteers 18.5 kg/m^2 ≤ BMI < 30 kg/m^2, weight(men) ≥55kg / weight(women) ≥45kg
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP <90 mmHg
* agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm or eggs from the date of administration of the first investigational drug to 7 days after the administration of the last investigational drug.
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
AUCt | 0~24 hours
  Pharmacokinetic evaluation
Cmax | 0~24 hours
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf | 0~24 hours
  Pharmacokinetic evaluation
Tmax | 0~24 hours
  Pharmacokinetic evaluation
t1/2 | 0~24 hours
  Pharmacokinetic evaluation
CL/F | 0~24 hours
  Pharmacokinetic evaluation
Vd/F | 0~24 hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, MD, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea